CLINICAL TRIAL: NCT03430687
Title: A Phase I Study of Intravesical Talimogene Laherparepvec for Non-Muscle Invasive Transitional Cell Carcinoma
Brief Title: Talimogene Laherparepvec in Treating Patients With Non-Muscle Invasive Bladder Transitional Cell Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigators prefer to pursue other studies
Sponsor: University of California, San Francisco (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15521; NCI-2018-00109 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-17558; 15521 (Other: UCSF Medical Center-Mount Zion)
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Stage 0 Bladder Urothelial Carcinoma AJCC v6 and v7; Stage 0a Bladder Urothelial Carcinoma AJCC v6 and v7; Stage 0is Bladder Urothelial Carcinoma AJCC v6 and v7; Stage I Bladder Urothelial Carcinoma AJCC v6 and v7
MeSH Terms: interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (talimogene laherparepvec) (Experimental): Patients receive talimogene laherparepvec intravesically (10ml of 10^6 PFU/mL) on days 1, 8, 15, 22, 29, and 36 or days 1, 15, and 29 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Talimogene Laherparepvec — Given intravesically
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase I trial studies the side effects and best dose of talimogene laherparepvec and to see how well it works in treating patients with non-muscle invasive bladder transitional cell carcinoma. Biological therapies, such as talimogene laherparepvec, use substances made from living organisms that may attack specific tumor cells and stop them from growing or kill them.

ELIGIBILITY:
Inclusion Criteria:

* Histologically document transitional cell carcinoma with the presence of any of the following stages: carcinoma in situ (CIS), high-grade Ta, or any grade T1, detectable at the time of study accrual; combinations of the aforementioned stages are acceptable; subjects with mixed histology are required to have a dominant transitional cell carcinoma (TCC) pattern
* Failure of prior intravesical treatment(s), one of which must include a course of BCG; failure is defined as evidence of TCC on cystoscopic examination and biopsy or cystoscopic examination and urine cytology at least 6 weeks from completion of last treatment
* Patient is either ineligible for or declines radical cystectomy; the investigator must explain that a delay in cystectomy may increase the patient?s chance of disease progression
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Ability to understand and willingness to sign written informed consent
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2.5 x institutional upper limit of normal (ULN) and total bilirubin < 1.5 x institutional ULN
* Absolut neutrophil count (ANC) > 1500/uL
* Platelets >= 75,000/uL
* Hemoglobin > 8 mg/dL without need for hematopoetic growth factor or transfusion support
* Estimated glomerular filtration rate (GFR) > 30 ml/min
* Serum creatinine less than 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance = or 60 mL/min for subject with creatinine levels more than 1.5 x ULN; (Note: creatinine clearance need not be determined if the baseline serum creatinine is within normal limits; creatinine clearance should be determined per institutional standard)
* Prothrombin time (PT)/international normalized ratio (INR), partial thromboplastin time (PTT) =< 1.5 x ULN
* No known history of human immunodeficiency virus (HIV) 1/2, human T-lymphotropic virus (HTLV)-I/II
* No currently active hepatitis B or C
* Males with partners of childbearing potential, must agree for the duration of the treatment with talimogene laherparepvec and continuing for 3 months after the last tumor injection of talimogene laherparepvec to either:

  * Abstain from sexual activity
  * Use highly effective barrier protection (latex condom)
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment; if urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * If a pregnancy occurs, the study doctor must be notified; the study doctor should notify the study sponsor as well as Amgen of the pregnancy, discuss any follow-up with the subject (and/or his partner), and ask for information on the pregnancy outcome; the patient should be asked if she wishes to consent to follow up through the Amgen pregnancy surveillance program
  * If the female partner is already pregnant when the male subject begins treatment with talimogene laherparepvec, he must refrain from any sort of sexual activity that could expose his partner or the unborn baby to talimogene laherparepvec through semen, or wear a latex condom during sexual activity while receiving treatment with talimogene laherparepvec and for at least 3 months after the last talimogene laherparepvec administration

Exclusion Criteria:

* Any subjects with muscle-invasive TCC (stages T2 - T4) OR any known TCC of the ureter or renal pelvis are not allowed
* Any history of metastatic TCC; subjects with suspected malignant lymphadenopathy in the abdomen or pelvis are not allowed
* Known active central nervous system (CNS) metastases; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids > 10 mg/day of prednisone or equivalent; the exception does not include carcinomatosus meningitis which is excluded regardless of clinical stability
* Patients whom, in the opinion of the treating urologic oncologist, should undergo cystectomy due to high-risk features
* Intravesical chemo- or biologic therapy within 6 weeks of first treatment
* Prior systemic chemotherapy for transitional cell carcinoma of the bladder; subjects who have received prior intravesical chemotherapy are allowed if completed 28 days prior to cycle 1 day
* Prior radiation therapy for TCC
* History or evidence of active autoimmune disease, requiring systemic steroid therapy within 28 days of study screening or other systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients on inhaled or topical steroids are eligible
  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the principal investigator
  * Replacement therapy (e.g., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Major surgery (requiring the use of a general anesthetic) within 4 weeks of study enrollment with the exception of transurethral resection of bladder tumor (TURBT)
* Concurrent use of investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec
* Malignancies other than urothelial cancer (UC) within 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent and absence of PSA relapse, or ductal carcinoma in situ of the breast treated surgically with curative intent) or incidental prostate cancer

  * Patients are considered to be free of active malignancy if they have completed therapy and have a < 30% risk of relapse
* Uncontrolled cystitis, gross hematuria, bladder pain, or bladder spasms, other uncontrolled concurrent illness, or any underlying medical condition, including any underlying conditions resulting in chronic immunosuppression which in the Investigator?s opinion will make the administration of talimogene laherparepvec hazardous, or obscure the interpretation of adverse events
* Currently known active infection with HIV, hepatitis B or C virus
* Clinically significant obstructive airway disease
* Active HSV infection requiring treatment, or requiring intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g. acyclovir)
* Pregnant or nursing women are excluded
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec
* Received live vaccine within 28 days prior to enrollment
* Active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis)
* Previous treatment with talimogene laherparepvec or any other oncolytic virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related toxicities according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (Dose escalation) | Up to 2 years
  The distribution for the maximum observed grade for each adverse event will be tabulated and reported with 95% confidence interval.
Pathologic T0 rate (Dose expansion) | At 6 months
  Point estimates and 95% confidence intervals will be obtained for each dose level of talimogene laherparepvec. Will be estimated for the expansion cohort and compared with the null hypothesis rate separately by using one-sample proportion test.
Relapse-free survival rate (Dose expansion) | From study start until recurrence of disease or death from any cause, assessed at 2 years
  Point estimates and 95% confidence intervals will be obtained for each dose level of talimogene laherparepvec. Will be estimated for the expansion cohort and compared with the null hypothesis rate separately by using one-sample proportion test.

SECONDARY OUTCOMES:
Change in antigen presenting cell (APC) within bladder tumor tissue by immunohistochemical (IHC) assessment | Baseline up to 2 years
  APC infiltration (CD68+, CD11c+, or CD83+) will be assessed by IHC staining, and quantitated by the number of APCs/um^2. Therefore, the number of APCs will be normalized per unit area. APC will be enumerated from 3 tissue regions: tumor/benign tissue interface (from here on referred to as the ?tumor interface?), tumor center, and benign glands
Change in circulating immune cells following intravesical talimogene laherparepvec, by flow cytometric assessment | Baseline up to 2 years
  Flow cytometry will be performed in both pre- and post-treatment peripheral blood mononuclear cells to determine the change in T cell activation (both regulatory T cells and T effector cells) after intravesical talimogene laherparepvec therapy. Descriptive statistics for continuous measurements will be used to summarize the changes.
Change in T cell and other immune cell infiltration within bladder tumor tissue by IHC assessment | Baseline up to 2 years
  T cell tumor infiltration (of selected T cell subsets) will be scored by IHC assessment, and scored by the number of T cells/um^2. Therefore, the number of T cells will be normalized per unit area. T cell-infiltration for both the pre- treatment diagnostic biopsy specimen and the post-treatment specimen will be quantitated in this fashion. Separate scores will be reported for further characterization of T cell infiltration for tumor interface, tumor center, and benign tissue.
Herpes simplex virus (HSV) status assessed by rate of HSV seroconversion in patients who were previously HSV-seronegative and relationship between HSV status and immunologic infiltration within tumor | Up to day 43
  In patients who were previously HSV-seronegative, the proportion of patients with HSV seroconversion will be reported, with 95% confidence intervals. The relationship between APC infiltration and baseline HSV status will be reported as a binary outcome: positive or negative. Patients with baseline HSV negative status who experience seroconversion will be assessed by the chi-square test separately.
Viral replication as measured by viral titers | Up to 2 years
  Viral replication will be assessed by urinary viral titers drawn and assessed by polymerase chain reaction and cellular based assays as previously described. These assays will be performed prior to each dose, as well as at +1 hour (h), +2 h, +24 h and +168 h, with a window of 6 hours for the +24 and +168 h to accommodate for logistical issues patients returning to the clinic. Results will be summarized descriptively as change from baseline using appropriate statistical methods.

OTHER OUTCOMES:
Antibody responses measured by spotted antigen arrays | Up to 6 weeks following therapy
  To characterize antibody responses to a broad panel of antigens, sera will be collected at baseline and 6 weeks following therapy, and profiled using spotted antigen array. After standard preprocess of the protein array data, Cluster and Treeview software will be used for unsupervised clustering of the data with Pearson correlation and complete linkage. For each array, an antigen is identified as being detected if its value is above the median. To determine the number of up- and down modulated antibodies, the difference in log2 intensity values of pretreatment and posttreatment samples will be
Apoptosis by IHC assessment of cleaved caspase-3 | Up to 2 years
  Will be scored on a 0-100 continuous scale based on % area that is positive for stain in regions of tumor. Special attention will be paid to areas of high grade tumor for scoring purposes; areas of interface, benign, and tumor tissue will be scored separately. For each subject, the change in cleaved caspase-3 IHC score following talimogene laherparepvec will be calculated in order to characterize the biological impact of talimogene laherparepvec in NMIBC. Descriptive statistics for continuous measurements will be used to summary the IHC score change for each location. Furthermore, univariate a
Change in PD-L1 expression by IHC assessment | Baseline up to 2 years
  For each subject, the change in PD-L1 expression score defined as either an increase of decrease by at least 1 (on a scale of 1-3) following talimogene laherparepvec will be calculated for exploratory characterization of the impact on PD-L1 expression of talimogene laherparepvec in non-muscle invasive bladder cancer. Descriptive statistics for categorical measurements will be used to summary the PD-L1 expression change for each location. Furthermore, univariate analysis (proportion test) will be applied to explore the PD-L1 expression score change between locations.
Pyroptosis by IHC assessment of cleaved caspace-1 | Up to 2 years
  Will be scored on a 0-100 continuous scale based on % area that is positive for stain in regions of tumor. Special attention will be paid to areas of high grade tumor for scoring purposes; areas of interface, benign, and tumor tissue will be scored separately. For each subject, the change in cleaved caspace-1 IHC score following talimogene laherparepvec will be calculated in order to characterize the biological impact of talimogene laherparepvec in NMIBC. Descriptive statistics for continuous measurements will be used to summary the IHC score change for each location. Furthermore, univariate a
T cell receptor deep sequencing of tissue samples from pre-treatment biopsies | Up to 2 years
T cell receptor deep sequencing of tissue samples from post-treatment resected tissues | Up to 2 years
T cell responses to candidate antigens measured by IFNgamma enzyme-linked immunosorbent spot assay | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Terence Friedlander, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States